CLINICAL TRIAL: NCT00879970
Title: AVANDIA CV Outcomes Study: Thiazolidinedione Intervention With Vitamin D Evaluation (TIDE) A Multicenter Randomized Double-Blind Placebo-Controlled Trial of a Thiazolidinedione or Placebo and of Vitamin D or Placebo In People With Type 2 Diabetes at Risk For Cardiovascular Disease
Brief Title: Thiazolidinedione Intervention With Vitamin D Evaluation
Acronym: TIDE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: FDA has placed the trial on full clinical hold.
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 111960
Record Dates: First submitted 2009-04-02; First posted 2009-04-13 (Estimated); Results first posted 2011-12-13 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Cardiovascular Outcomes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone; Rosiglitazone; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- pioglitazone (Active Comparator): PIO tablet was administered in the dose of 30 milligrams (mg) OD initially and could be titrated to a maximum dose of 45 mg at or after the 6-month visit. After 1 year of treatment, the dose of PIO was increased to 45 mg OD for the duration of 5.5 years.
  Interventions: Drug: pioglitazone
- rosiglitazone (Active Comparator): RSG tablet was administered in the dose of 4 mg OD initially and could be titrated to a maximum dose of 8 mg at or after the 6-month visit. After 1 year of treatment, the dose of RSG was increased to 8 mg OD for the duration of 5.5 years.
  Interventions: Drug: rosiglitazone
- TZD placebo (Placebo Comparator): Matching placebo tablet was administered once a day (OD) for the duration of 5.5 years
  Interventions: Drug: placebo
- Vitamin D (Active Comparator): Active comparator
  Interventions: Dietary Supplement: Vitamin D
- Vitamin D placebo (Placebo Comparator): Placebo Comparator
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Drug: pioglitazone — Pioglitazone30 mg and 45 mg tablets are over-encapsulated with Swedish orange size DB-AA capsule shell.
  Arms: pioglitazone
Drug: rosiglitazone — Rosiglitazone 4 mg and 8 mg tablets are over-encapsulated with Swedish orange size DB-AA capsule shell.
  Arms: rosiglitazone
Drug: placebo — Placebo to match is Swedish orange size DB-AA capsule filled with white to off-white non-active powder blend.
  Arms: TZD placebo
Dietary Supplement: Vitamin D — Vitamin D factor intervention
  Arms: Vitamin D
Dietary Supplement: Placebo — Vitamin D factor intervention
  Arms: Vitamin D placebo

SUMMARY:
This study will answer two separate questions.

The first question is to test the cardiovascular effects of long-term treatment with rosiglitazone or pioglitazone when used as part of standard of care compared to similar standard of care without rosiglitazone or pioglitazone in patients with type 2 diabetes who have a history of or are at risk for cardiovascular disease.

The second question will compare the effects of long-term supplementation of vitamin D on death and cancer

ELIGIBILITY:
Inclusion Criteria:

* Men or women with: a) newly detected type 2 diabetes based on a fasting plasma glucose greater than or equal to 7.0 mmol/l (126 mg/dL) or a 2 hour plasma glucose (FPG) greater than or equal to 11.1 mmol/l (200 mg/dL) on an oral glucose tolerance test, or b) a history of type 2 diabetes
* Hemoglobin A1c (A1C) 6.5-9.5% inclusive (for assays with upper limit of normal of 6%) within one month of screening
* Age ≥ 50 years and evidence of vascular disease defined as ≥1of:

  * prior myocardial infarction
  * prior stroke
  * coronary, carotid or peripheral artery revascularization ≥ 4 years earlier
  * previous documented myocardial ischemia on either an exercise stress test or on any cardiac imaging, or previous unstable angina with ECG changes or cardiac enzyme elevation OR
* Age ≥ 55 years and evidence of subclinical vascular disease defined as ≥1 of:

  * microalbuminuria or proteinuria
  * history of treated or untreated hypertension with left ventricular hypertrophy by electrocardiogram (ECG) or echocardiogram

    * 50% stenosis on any imaging of coronary, carotid or lower extremity arteries
  * ankle/brachial index <0.9 OR
* Age ≥ 60 years and at least 2 of the following cardiovascular disease risk factors:

  * current tobacco use
  * LDL-c ≥3.4 mmol/L (130 mg/dL) or on a lipid lowering medication
  * HDL-c < 1.0 mmol/L (40 mg/dL) for men and < 1.3 mmol/L (50 mg/dL) for women or triglycerides ≥ 2.3 mmol/L (200 mg/dL)
  * BP lowering medication use or untreated SBP ≥ 140 mmHg or DBP ≥ 95 mmHg
  * Waist to hip ratio > 1.0 for men and > 0.8 for women
* On no insulin and on less than or equal to 2 anti-diabetes drugs where at least one drug is at or below the half-maximal dose (as indicated in the MOP) with stable dosing for 10 weeks prior to screening

Exclusion Criteria:

* Type 1 diabetes
* Current need for insulin treatment
* Symptomatic hyperglycemia requiring immediate therapy in the judgment of the physician
* An acute cardiovascular event within 30 days prior to randomization
* Symptomatic heart failure (i.e. New York Heart Association class II or higher) or any episode of previous pulmonary edema or known ejection fraction < 0.4 or current use of loop diuretics
* Any fracture within the past 1 year
* Currently planned coronary, carotid or peripheral artery revascularization or cardiac valve surgery
* Coronary, carotid or peripheral artery revascularization within the 4 years prior to screening in the absence of angina, MI, or stroke in the intervening period
* End stage renal disease requiring renal replacement therapy
* Receiving drug therapy to treat liver disease
* A diagnosis of cancer (other than superficial squamous, basal cell skin cancer, or adequately treated cervical carcinoma in situ) in the past 3 years or current treatment for the active cancer (other than prophylactic)
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level > 2.5 times the upper limit of normal
* A prior heart transplant or awaiting a heart transplant
* Previous or current hypercalcemia, hyperparathyroidism, osteomalacia or other contraindication for vitamin D therapy
* Regular use of or indication for greater than 400IU of vitamin D daily
* Clinically or medically unstable with expected survival < 1 year
* Unwillingness to permit sites to contact their primary physicians to communicate information about the study and the participant's data
* Any other factor likely to limit protocol compliance or reporting of adverse events
* Inability to discontinue a TZD (if taking one) in the judgement of the physician/investigator
* Contraindications to or history of hypersensitivity to the investigational products
* History of renal stones within the past 2 years
* Participation in another clinical trial of an investigational agent

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1332 (Actual)
Dates: Start 2009-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (258):
- United States (22):
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Northridge, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Tucker, Georgia
  - GSK Investigational Site, Pocatella, Idaho
  - GSK Investigational Site, Pocatello, Idaho
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Haverhill, Massachusetts
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Kalispell, Montana
  - GSK Investigational Site, Westfield, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Temple, Texas
- Argentina (8):
  - GSK Investigational Site, Buenos Aires, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Coronel Suárez, Buenos Aires
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, San Nicolás de los Arroyos, Buenos Aires
  - GSK Investigational Site, Salta
  - GSK Investigational Site, San Miguel de Tucumán
  - GSK Investigational Site, Zárate
- Canada (25):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Surrey, British Columbia
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, St. John's, Newfoundland and Labrador
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Barrie, Ontario
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Cambridge, Ontario
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Ohsweken, Ontario
  - GSK Investigational Site, Oshawa, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Thornhill, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Laval, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Rimouski, Quebec
  - GSK Investigational Site, Saint-Georges, Quebec
  - GSK Investigational Site, Sainte-Foy, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- Chile (5):
  - GSK Investigational Site, Temuco, Región de La Araucania
  - GSK Investigational Site, Santiago, Región Metro de Santiago
  - GSK Investigational Site, Osorno
  - GSK Investigational Site, Valdivia
  - GSK Investigational Site, Victoria
- Colombia (12):
  - GSK Investigational Site, Armenia
  - GSK Investigational Site, Barrangquilla
  - GSK Investigational Site, Barranquilla
  - GSK Investigational Site, Bogotac
  - GSK Investigational Site, Bogotá
  - GSK Investigational Site, Cali
  - GSK Investigational Site, Cartagena
  - GSK Investigational Site, Espinal
  - GSK Investigational Site, Floridablanca
  - GSK Investigational Site, Manizales
  - GSK Investigational Site, Medellín
  - GSK Investigational Site, Pereira
- Czechia (8):
  - GSK Investigational Site, Havířov
  - GSK Investigational Site, Jihlava
  - GSK Investigational Site, Městec Králové
  - GSK Investigational Site, Ostrava
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Příbram
  - GSK Investigational Site, Rakovník
  - GSK Investigational Site, Uherské Hradiště
- Denmark (9):
  - GSK Investigational Site, Aarhus N
  - GSK Investigational Site, Copenhagen
  - GSK Investigational Site, Frederiksberg
  - GSK Investigational Site, Glostrup Municipality
  - GSK Investigational Site, Hellerup
  - GSK Investigational Site, Herlev
  - GSK Investigational Site, København NV
  - GSK Investigational Site, Odense C
  - GSK Investigational Site, Viborg
- Finland (3):
  - GSK Investigational Site, Helsinski
  - GSK Investigational Site, Kuopio
  - GSK Investigational Site, Oulu
- Germany (42):
  - GSK Investigational Site, Deggingen, Baden-Wurttemberg
  - GSK Investigational Site, Villingen-Schwenningen, Baden-Wurttemberg
  - GSK Investigational Site, Wangen, Baden-Wurttemberg
  - GSK Investigational Site, Weinheim, Baden-Wurttemberg
  - GSK Investigational Site, Augsburg, Bavaria
  - GSK Investigational Site, Gars Am Inn, Bavaria
  - GSK Investigational Site, Haag, Bavaria
  - GSK Investigational Site, Künzing, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Vilshofen, Bavaria
  - GSK Investigational Site, Wallerfing, Bavaria
  - GSK Investigational Site, Angermünde, Brandenburg
  - GSK Investigational Site, Elsterwerda, Brandenburg
  - GSK Investigational Site, Potsdam, Brandenburg
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Großalmerode, Hesse
  - GSK Investigational Site, Kelkheim, Hesse
  - GSK Investigational Site, Winsen/Lohe, Lower Saxony
  - GSK Investigational Site, Bad Oeynhausen, North Rhine-Westphalia
  - GSK Investigational Site, Bergkamen, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Dorsten, North Rhine-Westphalia
  - GSK Investigational Site, Eschweiler, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Witten, North Rhine-Westphalia
  - GSK Investigational Site, Ingelheim, Rhineland-Palatinate
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Rhaunen, Rhineland-Palatinate
  - GSK Investigational Site, Neunkirchen, Saarland
  - GSK Investigational Site, Borna, Saxony
  - GSK Investigational Site, Delitzsch, Saxony
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzg, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Oschatz, Saxony
  - GSK Investigational Site, Pirna, Saxony
  - GSK Investigational Site, Köthen, Saxony-Anhalt
  - GSK Investigational Site, Schönebeck, Saxony-Anhalt
  - GSK Investigational Site, Wolmirstedt, Saxony-Anhalt
  - GSK Investigational Site, Zerbst, Saxony-Anhalt
  - GSK Investigational Site, Berlin, State of Berlin
- India (17):
  - GSK Investigational Site, Ahmedabad
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Banjara Hills PO, Hyderabad
  - GSK Investigational Site, Belagavi
  - GSK Investigational Site, Chennai
  - GSK Investigational Site, Hyderabad
  - GSK Investigational Site, Karnāl
  - GSK Investigational Site, Kerala
  - GSK Investigational Site, Kochi
  - GSK Investigational Site, Kottyam
  - GSK Investigational Site, Mumbai
  - GSK Investigational Site, Nashik
  - GSK Investigational Site, Nellore
  - GSK Investigational Site, Pune
  - GSK Investigational Site, Tamil Nadu
  - GSK Investigational Site, Trivandrum
  - GSK Investigational Site, Vijayawada
- Italy (4):
  - GSK Investigational Site, Milano (Milan), Lombardy
  - GSK Investigational Site, Sesto San Giovanni (MI), Lombardy
  - GSK Investigational Site, Pozzilli (IS), Molise
  - GSK Investigational Site, Chieri (Torino)
- Latvia (6):
  - GSK Investigational Site, Cēsis
  - GSK Investigational Site, Daugavpils
  - GSK Investigational Site, Jēkabpils
  - GSK Investigational Site, Liepāja
  - GSK Investigational Site, Riga
  - GSK Investigational Site, Tukums
- Mexico (8):
  - GSK Investigational Site, Tijuana, Baja California Norte
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Zapopan, Jalisco
  - GSK Investigational Site, Morelia, Michoacán
  - GSK Investigational Site, San Luis Potosí City, San Luis Potosí
  - GSK Investigational Site, Aguascalientes
  - GSK Investigational Site, Guadalajara
  - GSK Investigational Site, Tampico
- Netherlands (4):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Heerlen
  - GSK Investigational Site, Hoofddorp
  - GSK Investigational Site, Rotterdam
- Norway (8):
  - GSK Investigational Site, Bodø
  - GSK Investigational Site, Hoenefoss
  - GSK Investigational Site, Kløfta
  - GSK Investigational Site, Oslo
  - GSK Investigational Site, Skedsmokorset
  - GSK Investigational Site, Stavanger
  - GSK Investigational Site, Tromsø
  - GSK Investigational Site, Trondheim
- Pakistan (3):
  - GSK Investigational Site, Faisalabad
  - GSK Investigational Site, Islamabad
  - GSK Investigational Site, Lahore
- GSK Investigational Site, Arequipa, Arequipa, Peru
- GSK Investigational Site, Laoag, Philippines
- Romania (11):
  - GSK Investigational Site, Bacau
  - GSK Investigational Site, Baia Mare
  - GSK Investigational Site, Bistriţa
  - GSK Investigational Site, Brasov
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Buzău
  - GSK Investigational Site, Deva
  - GSK Investigational Site, Iași
  - GSK Investigational Site, Oradea
  - GSK Investigational Site, Piteşti
  - GSK Investigational Site, Sibiu
- Russia (22):
  - GSK Investigational Site, Arkhangelsk
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Ivanovo
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Kirov
  - GSK Investigational Site, Kursk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Nizhny Novgorod
  - GSK Investigational Site, Ryazan
  - GSK Investigational Site, Saint Pertersburg
  - GSK Investigational Site, Saint Petersberg
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Smolensk
  - GSK Investigational Site, St'Petersburg
  - GSK Investigational Site, Syktyvkar
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Vladivostok
  - GSK Investigational Site, Volgograd
  - GSK Investigational Site, Voronezh
  - GSK Investigational Site, Yaroslavl
- Slovakia (2):
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Nitra
- South Africa (17):
  - GSK Investigational Site, Port Elizabeth, Eastern Cape
  - GSK Investigational Site, Meyerspark, Gauteng
  - GSK Investigational Site, Parktown, Gauteng
  - GSK Investigational Site, Chatsworth, KwaZulu-Natal
  - GSK Investigational Site, Umhlanga, KwaZulu-Natal
  - GSK Investigational Site, Bellville
  - GSK Investigational Site, Benoni
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Durban
  - GSK Investigational Site, Newton
  - GSK Investigational Site, Observatory
  - GSK Investigational Site, Parktown
  - GSK Investigational Site, Pretoria
  - GSK Investigational Site, Somerset West
  - GSK Investigational Site, Soweto
  - GSK Investigational Site, Worcester
- Sweden (12):
  - GSK Investigational Site, Eksjö
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Härnösand
  - GSK Investigational Site, Karlshamn
  - GSK Investigational Site, Kristianstad
  - GSK Investigational Site, Ljungby
  - GSK Investigational Site, Malmo
  - GSK Investigational Site, Oskarshamn
  - GSK Investigational Site, Skene
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Vaxjo
  - GSK Investigational Site, Vällingby
- GSK Investigational Site, Bangkok, Thailand
- United Kingdom (7):
  - GSK Investigational Site, Bath, Somerset
  - GSK Investigational Site, Chippenham
  - GSK Investigational Site, Doncaster
  - GSK Investigational Site, Harrogate
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Punthakee Z, Bosch J, Gerstein HC. Setting the record straight on TIDE: a lost opportunity for patients with diabetes. Diabetologia. 2013 Sep;56(9):1884-7. doi: 10.1007/s00125-013-2959-0. Epub 2013 Jun 6. PMID 23740195
- [Derived] Punthakee Z, Bosch J, Dagenais G, Diaz R, Holman R, Probstfield J, Ramachandran A, Riddle M, Ryden LE, Zinman B, Afzal R, Yusuf S, Gerstein H; TIDE Trial Investigators. Design, history and results of the Thiazolidinedione Intervention with vitamin D Evaluation (TIDE) randomised controlled trial. Diabetologia. 2012 Jan;55(1):36-45. doi: 10.1007/s00125-011-2357-4. Epub 2011 Oct 29. PMID 22038523
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 111960 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111960 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111960 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111960 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111960 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111960 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111960 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1332 participants were included in the TZD randomization, and 1221 of 1332 participants were included in the Vitamin D randomization.
Pre-assignment Details: Randomization occurred subsequent to a 3-week rosiglitazone (RSG) and vitamin D Single-blind Run-in Phase to assess compliance and tolerability. Participants received an RSG tablet (4 milligrams [mg]) and a vitamin D tablet (1000 international units [IU]) once a day.
Groups:
- Placebo: Matching placebo tablet was administered once a day (OD) for a mean duration of 162 days.
- Pioglitazone (PIO): PIO tablet was administered in the dose of 30-45 milligrams (mg) OD for a mean duration of 162 days.
- Rosiglitazone (RSG): RSG tablet was administered in the dose of 4-8 mg OD for a mean duration of 162 days.
- Vitamin D Placebo: Vitamin D placebo administered for a mean duration of 162 days.
- Vitamin D: 1,000 IU/day administered for a mean duration of 162 days.
Period: Period 1 TZD Randomization
Arm/Group | Placebo | Pioglitazone (PIO) | Rosiglitazone (RSG) | Vitamin D Placebo | Vitamin D
Started | 541 | 392 | 399 | 0 | 0
Completed | 533 | 388 | 393 | 0 | 0
Not Completed | 8 | 4 | 6 | 0 | 0
Not completed — Refused to Attend Final Visit | 3 | 3 | 4 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 0
Not completed — Death | 2 | 1 | 0 | 0 | 0
Not completed — Final or Study Hold Visits Not Completed | 2 | 0 | 1 | 0 | 0
Period: Period 2 Vitamin D Randomization
Arm/Group | Placebo | Pioglitazone (PIO) | Rosiglitazone (RSG) | Vitamin D Placebo | Vitamin D
Started | 0 | 0 | 0 | 614 | 607
Completed | 0 | 0 | 0 | 610 | 600
Not Completed | 0 | 0 | 0 | 4 | 7
Not completed — Refused to Attend Final Visit | 0 | 0 | 0 | 2 | 6
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Pioglitazone (PIO) | Rosiglitazone (RSG) | Total
Number analyzed (Participants) | 541 | 392 | 399 | 1332
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.4 (6.8) | 66.3 (6.6) | 66.5 (6.4) | 66.4 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 220 | 167 | 161 | 548
  Male | 321 | 225 | 238 | 784
Race/Ethnicity, Customized [Number; unit: participants]
  European/ Caucasian/ White | 330 | 241 | 255 | 826
  Unknown | 53 | 34 | 35 | 122
  South Asian | 63 | 46 | 48 | 157
  Black African | 45 | 35 | 26 | 106
  Native South American | 33 | 26 | 24 | 83
  Other Asian | 10 | 6 | 6 | 22
  Native North American | 1 | 2 | 4 | 7
  Japanese | 1 | 0 | 1 | 2
  Arab/ Persian | 1 | 1 | 0 | 2
  Native Hawaiian/ Australian or Other Asian Pacific | 1 | 1 | 0 | 2
  Malays | 1 | 0 | 0 | 1
  Sub-Saharan African | 1 | 0 | 0 | 1
  Missing | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Indicated Components of the Composite Cardiovascular Outcome for Thiazolidinedione (TZD)
Description: An event adjudication committee (EAC) adjudicated all occurrences of the components of the composite cardiovascular (CV; related to heart) outcome for TZD. Components are the first occurrence of cardiovascular death for which a non-heart-related cause has not been identified; non-fatal myocardial infarction (MI) (death of heart muscle from sudden blockage of a coronary artery by blood clot not leading to death); and non-fatal stroke (rapidly developing loss of brain function[s] due to disturbance in the blood supply to the brain not leading to death).
Time Frame: From Randomization at Visit 3 up to the Final Visit (average of 162 days)
Population: Intent-to-Treat (ITT) Population: all randomized participants
Measure: Number; unit: participants
Arm/Group | Placebo | Pioglitazone (PIO) | Rosiglitazone (RSG) | Vitamin D Placebo | Vitamin D
Number analyzed (Participants) | 541 | 392 | 399 | 614 | 607
participants
  CV Death/Non-Fatal MI/Non-Fatal Stroke | 5 | 2 | 1 | 3 | 2
  CV Death | 1 | 0 | 0 | 1 | 0
  Non-Fatal MI | 2 | 0 | 1 | 1 | 1
  Non-Fatal Stroke | 2 | 2 | 0 | 1 | 1

2. Primary Outcome: Number of Participants With the Indicated Components of the Composite Outcome for Vitamin D
Description: An EAC adjudicated all occurrences of the components of the composite outcome for vitamin D. Components are the first occurrence of death or cancer requiring hospitalization, treatment with medicines (chemotherapy), or surgery.
Time Frame: From Randomization at Visit 3 to Final Visit (up to 162 days)
Population: ITT Population
Measure: Number; unit: participants
Groups:
- Placebo: PLACEBO Matching placebo tablet was administered once a day (OD) for a mean duration of 162 days.
- Pioglitzaone: PIO tablet was administered in the dose of 30-45 milligrams (mg) OD for a mean duration of 162 days.
- Rosiglitazone: RSG tablet was administered in the dose of 4-8 mg OD for a mean duration of 162 days.
Arm/Group | Placebo | Pioglitzaone | Rosiglitazone | Vitamin D Placebo | Vitamin D
Number analyzed (Participants) | 541 | 392 | 399 | 614 | 607
participants
  Death or serious cancer | 6 | 3 | 1 | 3 | 2
  All death | 4 | 1 | 1 | 2 | 0
  Serious cancer | 2 | 2 | 0 | 1 | 2

3. Secondary Outcome: Number of Participants With Any Revascularization
Description: Revascularization is defined as any surgical procedure for the provision of a new, additional, or augmented blood supply to heart muscle. Data regarding the need for any revascularization were adjudicated by the EAC and sent to the data monitoring committee (IDMC) on a regular basis for unblinded review.
Time Frame: From Randomization at Visit 3 to Final Visit (up to 162 days)
Population: ITT Population
Measure: Number; unit: participants
Groups:
- Pioglitazone: PIO tablet was administered in the dose of 30-45 milligrams (mg) OD for a mean duration of 162 days.
Arm/Group | Placebo | Pioglitazone | Rosiglitazone | VITAMIN D PLACEBO | VITAMIN D
Number analyzed (Participants) | 541 | 392 | 399 | 614 | 607
participants | 6 | 3 | 5 | 7 | 5

4. Secondary Outcome: Number of Participants With Need for Hospitalization for Any Reason
Description: Data regarding the need for hospitalization for any reason were collected and were then forwarded to the independent data monitoring committee (IDMC) on a regular basis for unblinded review.
Time Frame: From Randomization at Visit 3 to Final Visit (up to 162 days)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | Pioglitazone | Rosiglitazone | VITAMIN D PLACEBO | VITAMIN D
Number analyzed (Participants) | 541 | 392 | 399 | 614 | 607
participants | 31 | 16 | 24 | 19 | 32

5. Secondary Outcome: Number of Participants With Need for Hospitalization for Congestive Heart Failure (CHF), Shortness of Breath, Pneumonia, or Angina
Description: CHF is a condition in which the heart is not able to pump adequate blood to meet the body's needs. Shortness of breath is defined as difficulty in breathing. Pneumonia is an infection of the lungs, caused by various microorganisms. Angina is defined as severe chest pain due to lack of adequate blood supply of the heart muscle because of obstruction/spasm of the heart's blood vessels. Data regarding the need for hospitalization due to any of these reasons were adjudicated by the EAC and sent to the IDMC on a regular basis for unblinded review.
Time Frame: From Randomization at Visit 3 to Final Visit (up to 162 days)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | Pioglitazone | Rosiglitazone | VITAMIN D PLACEBO | VITAMIN D
Number analyzed (Participants) | 541 | 392 | 399 | 614 | 607
participants
  CHF | 1 | 2 | 0 | 0 | 2
  Shortness of breath | 0 | 1 | 2 | 0 | 1
  Pneumonia | 0 | 1 | 0 | 0 | 0
  Angina | 3 | 1 | 1 | NA — Angina was not analyzed in the Vitamin D arm. | NA — Angina was not analyzed in the Vitamin D arm.

6. Secondary Outcome: Number of Participants With Composite Microvascular Outcome
Description: The components of the composite microvascular outcome are retinopathy, decline in eGFR, vitrectomy, and renal replacement surgery. Retinopathy is defined as damage to the inner lining of the eye (retina). Decline in eGFR is defined as a >=30% reduction in kidney function. Vitrectomy is a surgery to remove some or all of the fluid (vitreous humor) from the eye. Renal replacement therapy includes all the life-supporting treatments for renal failure. Data regarding the number of participants with changes in micro blood vessels (composite microvascular outcome) were collected at each visit.
Time Frame: From Randomization at Visit 3 to Final Visit (up to 162 days)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | Pioglitazone | Rosiglitazone | VITAMIN D PLACEBO | VITAMIN D
Number analyzed (Participants) | 541 | 392 | 399 | 614 | 607
participants | 21 | 8 | 9 | 18 | 18

7. Secondary Outcome: Number of Participants With Retinopathy Requiring Laser Therapy, a Decline in Estimated Glomerular Filtration Rate (eGFR), Vitrectomy, and Renal Replacement Therapy
Description: Retinopathy is defined as damage to the inner lining of the eye (retina). Decline in eGFR is defined as a >=30% reduction in kidney function. Vitrectomy is a surgery to remove some or all of the fluid (vitreous humor) from the eye. Renal replacement therapy includes all the life-supporting treatments for renal failure. Data on the number of participants with all of these microvascular outcomes were collected at each visit. Data regarding the number of participants with these microvascular outcomes were adjudicated by the EAC and sent to the IDMC on a regular basis for unblinded review.
Time Frame: From Randomization at Visit 3 to Final Visit (up to 162 days)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | Pioglitazone | Rosiglitazone | VITAMIN D PLACEBO | VITAMIN D
Number analyzed (Participants) | 541 | 392 | 399 | 614 | 607
participants
  Retinopathy Requiring Laser Therapy | 1 | 0 | 0 | 0 | 0
  Decline in eGFR >=30% | 20 | 8 | 9 | 18 | 18
  Vitrectomy | 0 | 0 | 0 | 0 | 0
  Renal Replacement Therapy | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Severe Lower Than Normal Blood Glucose Level (Hypoglycemia)
Description: Severe hypoglycemia is defined as hypoglycemia requiring assistance from another person with either a documented plasma glucose <=36 mg/deciliter (2.0 millimole per liter [mmol/L]) or prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration. Hypoglycemia data were obtained from outcomes reported by the site. Data regarding hypoglycemia were adjudicated by the EAC and sent to the IDMC on a regular basis for unblinded review.
Time Frame: From Randomization at Visit 3 to Final Visit (up to 162 days)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | Pioglitazone | Rosiglitazone | VITAMIN D PLACEBO | VITAMIN D
Number analyzed (Participants) | 541 | 392 | 399 | 614 | 607
participants | 0 | 2 | 1 | 0 | 3

9. Secondary Outcome: Number of Participants With Clinical Proteinuria
Description: Clinical proteinuria is defined as a laboratory detection of urinary protein excretion > 0.5 grams (g) per 24 hours; spot urine analysis for albumin:creatinine ratio >=300 milligrams/g; timed urine collection for albumin excretion >=200 µg/minute or >=300 mg/24 hours. Clinical proteinuria data were obtained from outcomes reported by the site.
Time Frame: From Randomization at Visit 3 to Final Visit (up to 162 days)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | Pioglitazone | Rosiglitazone | VITAMIN D PLACEBO | VITAMIN D
Number analyzed (Participants) | 541 | 392 | 399 | 614 | 607
participants | 1 | 0 | 0 | NA — Proteinuria was not analyzed in the Vitamin D arm. | NA — Proteinuria was not analyzed in the Vitamin D arm.

10. Secondary Outcome: Number of Participants With a Fracture
Description: Fracture is defined as a medical condition in which there is a break in the continuity of the bone. Fractures are defined as those breaks that are self reported plus confirmed by an X-ray. Data regarding all occurrences of any fracture were adjudicated by the EAC and sent to the IDMC on a regular basis for unblinded review.
Time Frame: From Randomization at Visit 3 to Final Visit (up to 162 days)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | Pioglitazone | Rosiglitazone | VITAMIN D PLACEBO | VITAMIN D
Number analyzed (Participants) | 541 | 392 | 399 | 614 | 607
participants | 2 | 2 | 3 | 3 | 3

11. Secondary Outcome: Number of Participants With Hepatic Enzyme Increased or Abnormal Liver Function Tests
Description: Liver function tests are groups of clinical biochemistry laboratory blood assays designed to give information about the health of the liver. "Liver function test abnormal" and "hepatic enzyme increased" were obtained from adverse event data as reported by investigators based on the reference range of the reporting local laboratory methodology. The vitamin D arm was not analyzed for this outcome measure.
Time Frame: From Randomization at Visit 3 to Final Visit (up to 162 days)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | Pioglitazone | Rosiglitazone | VITAMIN D PLACEBO | VITAMIN D
Number analyzed (Participants) | 541 | 392 | 399 | 614 | 607
participants | 1 | 0 | 1 | NA — The vitamin D arm was not analyzed for this outcome measure. | NA — The vitamin D arm was not analyzed for this outcome measure.

12. Secondary Outcome: Number of Participants With Cognitive (Mental Processes) Decline (CD) From Baseline to the Year 2 Visit and the Final Visit
Description: CD is equivalent to a difference of >=1.5 units on the Digit Symbol Substitution Test (DSST) score. The DSST is a neuropsychological test sensitive to brain damage, a serious loss of cognitive ability, age, and depression. It consists of digit-symbol pairs, followed by a list of digits. Under each digit the participant was asked to write the corresponding symbol as quickly as possible. The number of correct symbols within the allowed time (90 or 120 seconds) was measured in units (one correct score equals one unit).
Time Frame: From Randomization at Visit 3 to Final Visit (up to 162 days)
Population: ITT Population. Study participation was placed on full clinical hold before data could be collected for this endpoint.
Arm/Group | Placebo | Pioglitazone | Rosiglitazone | VITAMIN D PLACEBO | VITAMIN D
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Erectile Dysfunction
Description: Erectile dysfunction (ED) is sexual dysfunction characterized by the inability to develop or maintain an erection of the penis during sexual performance. ED was assessed by using the International Index of Erectile Dysfunction (IIED) questionnaire. This standardized and validated 15-item self-evaluation scale provides pre- and post-treatment clinic evaluations of erectile and orgasmic function, sexual desire, satisfaction with sexual intercourse, and general satisfaction.
Time Frame: From Randomization at Visit 3 to Final Visit (up to 162 days)
Population: ITT Population. Study participation was placed on full clinical hold before data could be collected for this endpoint.
Arm/Group | Placebo | Pioglitazone | Rosiglitazone | VITAMIN D PLACEBO | VITAMIN D
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Mean Score on Euro-QoL (EQ)-5D
Description: Quality of life (QoL) was assessed by using the Euro-QoL (EQ)-5D, a short questionnaire used for measuring health-related QoL. The preference weights are elicited by asking participants to place hypothetical health states on a visual analogue scale from "0" to "1", whereby a score of "1" represents the best health state imaginable and "0" represents a health state equivalent to being dead. Negative states are those worse than being dead.
Time Frame: From Randomization at Visit 3 to Final Visit (up to 162 days)
Population: ITT Population. Study participation was placed on full clinical hold before data could be collected for this endpoint.
Arm/Group | Placebo | Pioglitazone | Rosiglitazone | VITAMIN D PLACEBO | VITAMIN D
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Mean Score on Montreal Cognitive Assessment (MoCA) Test, as an Assessment of Cognitive Function (CF)
Description: CF was assessed with the 30-point (pt) MoCA test, involving a short-term memory recall task (T) (5 pts), a clock-drawing T (3 pts), a 3-dimensional cube copy (1 pt), a trail-making B T (1 pt), a phonemic fluency T (1 pt), a 2-item verbal abstraction T (2 pts), an attention T (1 pt), a serial subtraction T (3 pts), digits forward/ backward (1 pt each), a 3-item confrontation naming T (3 pts), repetition of 2 syntactically complex sentences (2 pts), and orientation to time/ place (6 pts). A score of 26 or above is normal.
Time Frame: From Randomization at Visit 3 to Final Visit (up to 162 days)
Population: ITT Population. Study participation was placed on full clinical hold before data could be collected for this endpoint.
Arm/Group | Placebo | Pioglitazone | Rosiglitazone | VITAMIN D PLACEBO | VITAMIN D
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 162 days for the TZD arm; 130 days for the vitamin D arm
Description: Non-serious AE's were not analyzed including the Vitamin D Placebo and Vitamin D arms. As a result, data is presented as "0" participants at risk for both the Vitamin D Placebo and Vitamin D arms.
Arm/Group | Placebo | Pioglitazone | Rosiglitazone | Vitamin D Placebo | Vitamin D
Serious Adverse Events (participants affected / at risk) | 7/541 | 5/392 | 2/399 | 2/614 | 9/607
Other Adverse Events (participants affected / at risk) | 36/541 | 35/392 | 21/399 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=541) | Pioglitazone (N=392) | Rosiglitazone (N=399) | Vitamin D Placebo (N=614) | Vitamin D (N=607)
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 2
Angioplasty (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Aortic aneurysm repair (Surgical and medical procedures) | 1 | 0 | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1
Intestinal prolapse (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Multi-organ failure (General disorders) | 1 | 0 | 0 | 0 | 0
Pruritis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=541) | Pioglitazone (N=392) | Rosiglitazone (N=399) | Vitamin D Placebo (N=0) | Vitamin D (N=0)
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 3 | 2 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Right ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 3 | 1 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 3 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 2 | 0 | 0
Drug intolerance (General disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 0 | 0 | 0
Malaise (General disorders) | 1 | 3 | 0 | 0 | 0
Edema (General disorders) | 2 | 5 | 1 | 0 | 0
Edema peripheral (General disorders) | 4 | 8 | 1 | 0 | 0
Swelling (General disorders) | 1 | 0 | 0 | 0 | 0
Temperature intolerance (General disorders) | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cardiac stress test abnormal (Investigations) | 1 | 0 | 0 | 0 | 0
Catheterisation cardiac (Investigations) | 0 | 0 | 1 | 0 | 0
Echocardiogram abnormal (Investigations) | 1 | 0 | 0 | 0 | 0
Ejection fraction abnormal (Investigations) | 1 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Electrocardiogram abnormal (Investigations) | 1 | 0 | 0 | 0 | 0
Electrocardiogram change (Investigations) | 1 | 0 | 0 | 0 | 0
Glycosylated hemoglobin increased (Investigations) | 0 | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 2 | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Renal cancer (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Bladder obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 4 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin discoloration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Hospitalization (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Surgery (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The intended duration of this study was approximately 5.5 years. However, the trial was stopped prematurely because of regulatory concerns after a mean of 162 days without consideration of the accrued data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.